CLINICAL TRIAL: NCT01323244
Title: A Phase III, Open-Label, Single Arm, Rollover Trial of TMC435 in Combination With Peginterferon Alpha-2A and Ribavirin for HCV Genotype-1 Infected Subjects Who Participated in the Placebo Group of a Phase II/III TMC435 Study, or Who Received DAA Treatment in a Tibotec-Sponsored Phase I Study.
Brief Title: A Study of TMC435 in Combination With Peginterferon Alfa-2A and Ribavirin for Hepatitis C Virus Genotype-1 Infected Patients Who Participated in a Control Group of a TMC435 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017983; TMC435-TiDP16-C213 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C
Keywords: TMC435-TiDP16-C213; TMC435-C213; TMC435; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC435 (Experimental): TMC435 Type=exact number unit=mg number=150 form=capsule route=oral use once daily for 12 weeks in addition to peginterferon alfa-2a peginterferon and ribavirin for 24 or 48 weeks
  Interventions: Drug: TMC435

INTERVENTIONS:
Drug: TMC435 — Type=exact number, unit=mg, number=150, form=capsule, route=oral use, once daily for 12 weeks in addition to peginterferon alfa-2a peginterferon and ribavirin for 24 or 48 weeks

SUMMARY:
The purpose of this study is to investigate the efficacy of a treatment with TMC435 in combination with peginterferon alfa-2a and ribavirin in patients who did not clear their hepatitis C infection with peginterferon alfa-2a and ribavirin alone within a previous trial conducted by Tibotec, or who participated in Tibotec trials in which antivirals directed against hepatitis C virus (HCV) were evaluated for short periods of time.

DETAILED DESCRIPTION:
This is a roll over trial of TMC435 for patients with genotype-1 HCV infection who participated in the control (placebo; substance containing no active medication) group of a TMC435 trial or who received a treatment for up to 14 days with antivirals directed against HCV in a previous Tibotec trial. Patients in this study will receive TMC435 in combination with peginterferon alfa-2a (Pegasys) and ribavirin (Copegus) followed by peginterferon alfa-2a and ribavirin alone. The total treatment duration will be 24 or 48 weeks, depending on how the patients respond to treatment and which was their previous response to peginterferon alfa-2a and ribavirin alone. The study doctor will inform each patient about how to take their study medication and when they should stop taking it. After a patient stops taking study medication, they will contiue to come to the doctor's office for study visits until 24 weeks (in some cases up to 48 weeks) after end of treatment. The total duration of the study is 78 weeks (including screening). Patients will be monitored for safety throughout the study. Study assessments at each visit may include but are not limited to: blood and urine collection for testing, electrocardiogram (ECG) assessments (a measurement of the electrical activity of the heart) and physical examinations. TMC435 will be taken as an oral capsule of 150 mg once per day. Peginterferon (Pegasys) will be given as an injection of 180 µg once each week. Ribavirin will be taken as tablets (Copegus) twice each day and the dose will depend on patient's body weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the placebo arm of a TMC435 study who did not achieve undetectable HCV RNA levels at end of treatment or who relapsed within 1 year after end of treatment OR Patients who received short-term direct-acting antiviral therapy in a Tibotec-sponsored study.
* Liver disease stage documented by liver biopsy is required within 3 years prior to screening unless contraindicated.

Exclusion Criteria:

* Infection with human immunodeficiency virus.
* Liver disease not related to hepatitic C infection.
* Significant laboratory abnormalities or other active diseases.
* Pregnant or planning to become pregnant.
* Prematurely stopped medication in previous TMC435 study for non-compliance or for safety reasons.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with sustained viral response | 12 weeks after planned end of treatment

SECONDARY OUTCOMES:
The proportion of participants with sustained viral response | 24 weeks after planned end of treatment
Number of participants with HCV RNA level >1000 IU/mL | Week 4
Number of participants with viral breakthrough | Through Week 48
Number of participants with viral relapse | Through Week 48
Number of participants with normalized alanine aminotransferase levels | Through Week 48
Number of participants with on-treatment failure | Through Week 48
Number of participants affected by an adverse event | Through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (72):
- United States (15):
  - Bakersfield, California
  - Los Angeles, California
  - San Diego, California
  - Englewood, Colorado
  - Jacksonville, Florida
  - Orlando, Florida
  - New Orleans, Louisiana
  - Jackson, Mississippi
  - Tupelo, Mississippi
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
- Argentina (2):
  - Buenos Aires
  - Rosario, Santa Fe
- Australia (5):
  - Adelaide
  - Concord
  - Melbourne
  - Wentworthville
  - Woolloongabba
- Vienna, Austria
- Belgium (3):
  - Antwerp
  - Brussels
  - Ghent
- São Paulo, Brazil
- Sofia, Bulgaria
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- France (4):
  - Grenoble
  - Lyon
  - Nice Cedex 03 N/A
  - Paris
- Germany (7):
  - Berlin
  - Frankfurt A. M.
  - Hamburg
  - Kiel
  - Münster
  - Ulm
  - Würzburg
- Israel (2):
  - Haifa
  - Safed
- Monterrey, Mexico
- Netherlands (2):
  - Amsterdam
  - Rotterdam
- New Zealand (2):
  - Auckland
  - Christchurch
- Poland (6):
  - Bydgoszcz
  - Chorzów
  - Czeladź
  - Kielce
  - Mysłowice
  - Warsaw
- Portugal (2):
  - Coimbra
  - Lisbon
- San Juan, Puerto Rico
- Bucharest, Romania
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
- Spain (4):
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- Ukraine (3):
  - Donetsk
  - Kyiv
  - Vinnitsa
- United Kingdom (2):
  - Birmingham
  - London

REFERENCES:
- [Derived] Gane EJ, DeJesus E, Janczewska E, George J, Diago M, Da Silva MH, Reesink H, Nikitin I, Hinrichsen H, Bourgeois S, Ferenci P, Shukla U, Kalmeijer R, Lenz O, Fevery B, Corbett C, Beumont M, Jessner W. Simeprevir with peginterferon alpha-2a/ribavirin for chronic hepatitis C virus genotype 1 infection in treatment-experienced patients: an open-label, rollover study. BMC Infect Dis. 2017 Jun 2;17(1):389. doi: 10.1186/s12879-017-2444-3. PMID 28577353
- See also: A Study of TMC435 in Combination with Peginterferon Alfa-2A and Ribavirin for Hepatitis C Virus Genotype-1 Infected Patients who Participated in a Control Group of a TMC435 Study. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=1054&filename=CR017983_CSR.pdf